CLINICAL TRIAL: NCT01615822
Title: A Phase I Healthy Volunteer Study Investigating the Safety, Tolerability & Pharmacokinetics of Co-administered Single Doses of OZ439 and Mefloquine
Brief Title: Safety, Tolerability & Pharmacokinetics (PK) of Co-administered Single Doses of OZ439 and Mefloquine (MQ) in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision taken to halt progression of mefloquine as a potential partner for OZ439 as a single dose cure due to low probability of success
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMV_OZ439_12_001
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Malaria
Keywords: Malaria; PK; OZ439; Mefloquine; Healthy Volunteers
MeSH Terms: conditions — Malaria | interventions — artefenomel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- OZ439 100mg single dose (Experimental): OZ439 100mg single dose oral suspension
  Interventions: Drug: OZ439 100mg
- OZ439 100mg plus MQ 250mg single doses (Experimental): Single dose OZ439 100mg oral suspension in combination with single dose MQ 250mg tablet
  Interventions: Drug: OZ439 100mg; Drug: MQ 250 mg, single dose
- OZ439 400mg single dose (Experimental): OZ439 400mg single dose oral suspension
  Interventions: Drug: OZ439 400mg
- OZ439 400mg plus MQ 750mg single doses (Experimental): Single dose OZ439 400mg oral suspension in combination with single dose MQ 750mg tablets
  Interventions: Drug: OZ439 400mg; Drug: MQ 750mg, single dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OZ439 100mg — OZ439 100mg oral suspension, single dose
  Arms: OZ439 100mg plus MQ 250mg single doses; OZ439 100mg single dose
Drug: OZ439 400mg — OZ439 400mg oral suspension, single dose
  Arms: OZ439 400mg plus MQ 750mg single doses; OZ439 400mg single dose
Drug: MQ 250 mg, single dose — Mefloquine 250 mg tablet, single dose
  Arms: OZ439 100mg plus MQ 250mg single doses
Drug: MQ 750mg, single dose — Mefloquine 750mg oral tablet, single dose
  Arms: OZ439 400mg plus MQ 750mg single doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
OZ439 is a novel, synthetic trioxolane medicine which is related to artemisinin, but has the advantage of a longer elimination half-life so is being developed to be administered together with a potential partner drug e.g. mefloquine as a single dose cure for uncomplicated malaria. The study findings will be used to inform the dose and design of future studies. The aim of the study is to establish the safety, tolerability and pharmacokinetics of co-administered OZ439 and MQ at a range of doses up to the maximum tolerated dose, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-childbearing potential female volunteers of between 18 and 55 years of age
* Female volunteers must have a negative serum pregnancy test at screening
* Females must be of non-childbearing potential
* Male volunteers and their partner(s) must agree to use a double barrier method of contraception for at least 14 days prior to first dose of study drug through 90 days after the last dose.
* Body mass Index between 18 and 30kg/m2, inclusive; and a total body weight >50 kg
* Laboratory tests at screening within normal ranges or not clinically significant as judged by the Investigator.

Exclusion Criteria:

* Received an investigational drug or participated in another research study within 30 days of the first dose of study drug or at any time through the study
* Evidence of current or history of clinically significant oncologic, pulmonary, hepatic, cardiovascular, gastrointestinal, haematologic, metabolic, neurological, immunologic, nephrologic, endocrine, psychiatric disease, or clinically significant current infection.
* Any condition that could possibly affect drug absorption, such as gastrectomy, diarrhea and lactose intolerance
* Use of any medications, vitamins, herbal supplements, dietary supplements or vaccinations within 14 days of the first dose of study drug or at any time through the study, unless prior approval is granted. This includes any drugs that are substrates, inhibitors or inducers of CYP3A4. Intermittent use of acetaminophen at doses of up to 2g/day is permitted
* History of drug or alcohol abuse within 2 years of Screening
* History of alcohol consumption within 24 hours of any study visit
* Tobacco users
* Consumption of fruit juices within 7 days prior to dosing
* Participation in unaccustomed strenuous exercise within 7 days prior to
* Positive urine drug screen
* Positive test for HIV-1, HBsAg or HCV
* Known hypersensitivity to MQ or artemisinins
* QTcF greater than 450msec

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen I Barnes, Principal Investigator — University of Cape Town
Locations (1):
- Division of Clinical Pharmacology, University of Cape Town, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Period 1: OZ439 100mg single dose oral suspension
  Period 2: Single dose OZ439 100mg oral suspension in combination with single dose MQ 250mg tablet
- Cohort 2: Period 1: OZ439 400mg single dose oral suspension
  Period 2: Single dose OZ439 400mg oral suspension in combination with single dose MQ 750mg tablets
Period: Period 1
Arm/Group | Cohort 1 | Cohort 2 | Placebo
Started | 8 | 11 | 6
Completed | 7 | 9 | 6
Not Completed | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Period: Period 2
Arm/Group | Cohort 1 | Cohort 2 | Placebo
Started | 7 | 9 | 6
Completed | 7 | 8 | 4
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: In Cohort 2, one subject withdrew consent prior to dosing and is therefore not part of the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (10.3) | 30.6 (9.42) | 26 (4.45) | 28.6 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 7 | 8 | 6 | 21
Region of Enrollment [Number; unit: participants]
  South Africa | 8 | 10 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: OZ439 AUC0-t
Description: Area under the plasma concentration versus time curve (AUC) of OZ439
Time Frame: Up to 42 days post-dose
Population: Only the subjects who completed all treatments in their respective cohort (per-protocol set) were included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | OZ439 100mg Single Dose | OZ439 100mg Plus MQ 250mg Single Doses | OZ439 400mg Single Dose | OZ439 400mg Plus MQ 750mg Single Doses
Number analyzed (Participants) | 7 | 7 | 9 | 9
ng*h/mL | 1060 (32) | 1060 (32) | 8100 (30) | 7300 (30)

2. Secondary Outcome: OZ439 Cmax
Description: Peak Plasma Concentration (Cmax) of OZ439
Time Frame: Up to 42 days post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | OZ439 100mg Single Dose | OZ439 100mg Plus MQ 250mg Single Doses | OZ439 400mg Single Dose | OZ439 400mg Plus MQ 750mg Single Doses
Number analyzed (Participants) | 7 | 7 | 9 | 9
ng/mL | 157 (24) | 147 (33) | 821 (21) | 745 (26)

3. Secondary Outcome: MQ AUC0-t
Description: Area under the plasma concentration versus time curve (AUC) of MQ
Time Frame: Up to 42 days post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | OZ439 100mg Plus MQ 250mg Single Doses | OZ439 400mg Plus MQ 750mg Single Doses
Number analyzed (Participants) | 7 | 8
ng*h/mL | 167 (18) | 421 (30)

4. Secondary Outcome: MQ Cmax
Description: Peak Plasma Concentration (Cmax) of MQ
Time Frame: Up to 42 days post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | OZ439 100mg Plus MQ 250mg Single Doses | OZ439 400mg Plus MQ 750mg Single Doses
Number analyzed (Participants) | 7 | 8
ng/mL | 0.602 (27) | 1.34 (36)

ADVERSE EVENTS:
Time Frame: Up to Day 42 post-dose
Description: All subjects who received at least one dose of study drug were included in the safety analysis set. Adverse events were collected irrespective of whether or not the patients had received OZ439 alone or in combination with MQ.
Arm/Group | Cohort 1 | Cohort 2 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 9/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10) | Placebo (N=6)
Gun Shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Apart from a single gunshot wound, assessed as unrelated to investigational product, no other serious adverse events (SAEs) were reported
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=10) | Placebo (N=6)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical Device Site Reaction (General disorders) | 6 (6) | 6 (6) | 4 (4)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharynigitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea Cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional Arousal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depressive Symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Motion Sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ECG QT Shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
GGT Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No